CLINICAL TRIAL: NCT00721812
Title: A First Time In Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK1399686 After Single and Repeated Oral Dosing in Healthy Volunteers Using a Dose-Escalating, Randomized, Placebo-Controlled Study Design
Brief Title: A First Time In Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK1399686
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 111406
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: pharmacokinetics; Phase 1; first time in humans; IBD; safety; human volunteers
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A (Other): Single dose escalation
  Interventions: Drug: GSK1399686
- Part B (Other): 14 day repeat dose escalation
  Interventions: Drug: GSK1399686
- Part C (Other): Fixed dose food effect
  Interventions: Drug: GSK1399686

INTERVENTIONS:
Drug: GSK1399686 — Safety and tolerability dose escalation in normal human volunteers

SUMMARY:
A First-Time-in-Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of GSK1399686 After Single and Repeated Oral Dosing in Healthy Volunteers

ELIGIBILITY:
Inclusion criteria:

* Healthy as determined by a responsible physician
* Male, or only for the RDF cohort female of non-childbearing potential, between 18 and 65 years of age.
* Body weight greater than 50 kg (110 lbs) and BMI within the range 18.5-29.9 kg/m2 (inclusive).
* QTcB or QTcF < 450 msec
* Capable of giving written informed consent

Exclusion criteria:

* The subject has a positive pre-study drug/alcohol screen
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of greater than 21 units
* Urinary cotinine levels indicative of active smoking or regular use of tobacco
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody
* A positive test for HIV antibody
* The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives of the investigational product
* Exposure to more than four new chemical entities within 12 months
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices within 7 days
* Subject is receiving hormone replacement therapy
* History of sensitivity to any of the study medications
* History of sensitivity to heparin or heparin-induced thrombocytopenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-09-25 (Actual); Primary Completion 2009-05-27 (Actual); Study Completion 2009-05-27 (Actual)

PRIMARY OUTCOMES:
• Safety and tolerability as determined by AE reporting and treatment effects on vital signs, ECG findings, haematology, clinical chemistry and urinalysis parameters, as well as 24-hour plasma cortisol profiles | 72 hours and 14 days

SECONDARY OUTCOMES:
PK parameters per protocol | 72 hours and 14 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Harrow, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 111406 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111406?search=study&study_ids=111406#rs
- Available data/document: Clinical Study Report: 111406 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111406 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111406 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111406 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111406 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111406 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111406 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register